CLINICAL TRIAL: NCT03041766
Title: Safety and Immunogenicity Evaluation of the Vaccine Candidate Sm14 in Combination With the Adjuvant Glucopyranosyl Lipid A (GLA-SE) in Adults Living in Endemic Regions for S. Mansoni and S. Haematobium in Senegal. A Comparative, Randomized, Open-label Trial
Brief Title: Study of Safety and Immune Response of the Sm14 Vaccine in Adults of Endemic Regions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Orygen Biotecnologia SA (Unknown); Biomedical Research Center EPLS (Other); Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Principal Investigator, MIRIAM TENDLER, MD, PhD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sm14-2a-Sn
Record Dates: First submitted 2016-11-16; First posted 2017-02-03 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-01

CONDITIONS: Schistosomiasis
Keywords: Schistosomiasis; Recombinant vaccine; rSm14; GLA-SE; Fatty acid-binding protein (FABP); Phase II Clinical Trial; Senegal
MeSH Terms: conditions — Schistosomiasis | interventions — SM14 protein, Schistosoma mansoni; glucopyranosyl lipid-A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Adults with an infectious history of S. haematobium and S. mansoni and pretreated with 1 dose of Praziquantel (3 weeks prior to the first vaccine injection) receiving three (3) intramuscular injections of 50 μg Sm14 with 2.5 μg GLA-SE solution at D0, W4, W8 (D=day; W=week). Three-month follow-up (W12, W20).
  Interventions: Biological: Sm14; Drug: GLA-SE solution
- Group 2 (Experimental): Adults with an infectious history of S. haematobium and S. mansoni and pretreated with 1 dose of Praziquantel (3 weeks prior to the first vaccine injection) receiving three (3) intramuscular injections of 50 μg Sm14 with 5.0 μg GLA-SE solution at D0, W4, W8 (D=day; W=week). Three-month follow-up (W12, W20).
  Interventions: Biological: Sm14; Drug: GLA-SE solution

INTERVENTIONS:
Biological: Sm14 — Three 0.5 mL intra-muscular injections of the vaccine solution (50µg Sm14) will be administered on D0, W4, W8 (D = day, W = week).
  Other Names: rSm14
Drug: GLA-SE solution — Two (2) adjuvant concentrations will be made and packaged at 0.4 mL/vial, per GMP standards. One lot at the concentration of 10µg/mL for injection in the first cohort at 2.5µg GLA-SE/injection and one lot at the concentration of 20µg/mL for the second cohort intended to receive 5.0µg of GLA-SE/injection
  Other Names: Glucopyranosyl Lipid A in Stable Emulsion; Glucopyranosyl Lipid Adjuvant-Stable Emulsion; Toll-like Receptor 4 Agonist GLA-SE

SUMMARY:
The clinical trial phase 2a is designed to assess the safety of the active ingredient (protein + adjuvant) and secondarily its immunogenicity in healthy male adults from 18 to 49 years of age with a history of infection with intestinal and urinary schistosomiasis, living in the Valley of the Senegal River, a highly endemic area for schistosomiasis. Two arms in the study will test different doses of GLA-SE adjuvant (2.5 and 5 μg). This phase IIA in adults is considered to be a preliminary step in safety before starting trials in children in endemic areas to S. mansoni or S. haematobium, target population of the vaccine.

DETAILED DESCRIPTION:
A phase 2a trial, self-contained, open-label, randomized, dose-escalation study in two parallel arms receiving three (3) injections at D0, D28, D56; both groups receiving 50 μg Sm14 vaccine candidate solution, either combined with 2.5µg GLA-SE for the first group and 5µg for the second one in adults living in a S. mansoni and S. haematobium endemic area.

Sm14: recombinant protein produced in yeast following Good Manufacturing Practices (GMP) conditions, presented in vials containing 0.55 ml solution Sm14, 0.4 ml solution is diluted with 0.4 ml of GLA (Synthetic Glucopyranosyl lipid A) for intramuscular administration.

Medical examinations are performed at D0 (before injection, 1 hr and 4 hr after), and a safety evaluation at 24 hrs and 48 hrs, after each injection.

Blood analysis: Liver function tests - renal function tests - blood counts, at W-1 before inclusion, and then 7 days after each injections and at W13 and W21 during the follow-up.

Blood samples for immune response analysis at time of each injection, and then W12 and W20.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male, 18 to 49 years old (inclusive) at the time of inclusion.
* Living in one of selected villages in Saint-Louis Region (Senegal).
* Free of obvious/severe health problems except schistosomiasis, as established by clinical examination and blood analysis, i.e. hematological exams, liver and renal function tests.
* Written informed consent to participate obtained
* Treated with 40mg/kg Praziquantel (PZQ) before inclusion (W-5 to W-4 before the first injection) in case of infection with S. mansoni and S. haematobium
* Residence in the area during the period of the study.

Exclusion Criteria:

* Adult who does not respond to one of the inclusion criteria
* Current or previous chronic administration (defined as more than 14 days) of immunosuppressive drugs or other immuno-modifying drugs.
* Known hypersensitivity to any component in the Sm14 vaccine or history of allergic disease.
* Knowledge of non-infectious chronic disease
* Acute disease at time of enrollment.
* Other conditions which in opinion of the PI may potentially represent a danger for the patient to be enrolled.
* Non residence in the study area or intent to move during the study period

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability. | within 7 days of the administration of the first dose
  . Local signs and symptoms included Pain, Swelling and Inflammation at the injection site, Heaviness or pain upon passive or active movement of the injected limb, Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances. Laboratory tests (blood count, liver and kidney biological functions).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D30-D37: within 7 days of the administration of the second dose
  . Local signs and symptoms included Pain, Swelling and Inflammation at the injection site, Heaviness or pain upon passive or active movement of the injected limb, Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances. Laboratory tests (blood count, liver and kidney biological functions).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D60-67 : within 7 days of the administration of the third dose
  Local signs and symptoms included Pain, Swelling and Inflammation at the injection site. Heaviness or pain upon passive or active movement of the injected limb, Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances. Laboratory tests (blood count, liver and kidney biological functions).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D90 : three months after the first injection
  injection Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances. Laboratory tests (blood count, liver and kidney biological functions).
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | D120 : four months after the first injection
  Local signs and symptoms included pain or tenderness, swelling, induration and erythema at the site of injection. Complete physical examination including an examination of general appearance, body weight and forehead temperature, head, eyes, ears, nose and throat, neck, skin, cardiovascular and respiratory system, abdominal system, nervous system, lymphatic area, blood pressure, pulse and respiratory rates. General signs and symptoms including fever, headache, nausea, vomiting, myalgia, arthralgia, irritability/fussiness and drowsiness, loss of appetite and sleep disturbances. Laboratory tests (blood count, liver and kidney biological functions).

SECONDARY OUTCOMES:
Qualitative and quantitative assessment of the Immunogenicity | Day of first administration
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).
Qualitative and quantitative assessment of the Immunogenicity | 30 days after the first administration
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).
Qualitative and quantitative assessment of the Immunogenicity | 60 days after the first administration
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).
Qualitative and quantitative assessment of the Immunogenicity | 90 days after the first administration
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).
Qualitative and quantitative assessment of the Immunogenicity | 120 days after the first administration
  Immunogenicity was evaluated by Isotype analysis of the antibodies produced specifically against the rSm14 and vaccine-induced (ELISA) and Specific rSm14 cellular response (on PBMC), production of intracellular cytokines (PBMCs stimulation and cytokine dosing). Cellular immune responses measured by PBMC luminex assay for T-cell cytokines (Milliplex ® MAP kit).
  Correlation between the development and magnitude of humoral responses measured by antibody IgG production to the Sm14 Schisto protein using enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Tendler, MD, PhD, Study Chair — Oswaldo Cruz Foundation; Doudou DIOP, MD, Principal Investigator — Biomedical Research Center ESPOIR POUR LA SANTE (BRC-EPLS); Gilles RIVEAU, PharmD, PhD, Study Director — Biomedical Research Center ESPOIR POUR LA SANTE (BRC-EPLS)
Locations (1):
- Biomedical Research Center EPLS, Saint-Louis, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moser D, Tendler M, Griffiths G, Klinkert MQ. A 14-kDa Schistosoma mansoni polypeptide is homologous to a gene family of fatty acid binding proteins. J Biol Chem. 1991 May 5;266(13):8447-54. PMID 2022660
- [Result] Ramos CR, Spisni A, Oyama S Jr, Sforca ML, Ramos HR, Vilar MM, Alves AC, Figueredo RC, Tendler M, Zanchin NI, Pertinhez TA, Ho PL. Stability improvement of the fatty acid binding protein Sm14 from S. mansoni by Cys replacement: structural and functional characterization of a vaccine candidate. Biochim Biophys Acta. 2009 Apr;1794(4):655-62. doi: 10.1016/j.bbapap.2008.12.010. Epub 2008 Dec 25. PMID 19150418
- [Result] Coler RN, Bertholet S, Moutaftsi M, Guderian JA, Windish HP, Baldwin SL, Laughlin EM, Duthie MS, Fox CB, Carter D, Friede M, Vedvick TS, Reed SG. Development and characterization of synthetic glucopyranosyl lipid adjuvant system as a vaccine adjuvant. PLoS One. 2011 Jan 26;6(1):e16333. doi: 10.1371/journal.pone.0016333. PMID 21298114
- [Result] Santini-Oliveira M, Coler RN, Parra J, Veloso V, Jayashankar L, Pinto PM, Ciol MA, Bergquist R, Reed SG, Tendler M. Schistosomiasis vaccine candidate Sm14/GLA-SE: Phase 1 safety and immunogenicity clinical trial in healthy, male adults. Vaccine. 2016 Jan 20;34(4):586-594. doi: 10.1016/j.vaccine.2015.10.027. Epub 2015 Nov 10. PMID 26571311
- [Result] Lambert SL, Yang CF, Liu Z, Sweetwood R, Zhao J, Cheng L, Jin H, Woo J. Molecular and cellular response profiles induced by the TLR4 agonist-based adjuvant Glucopyranosyl Lipid A. PLoS One. 2012;7(12):e51618. doi: 10.1371/journal.pone.0051618. Epub 2012 Dec 28. PMID 23284726